CLINICAL TRIAL: NCT02479191
Title: The LUCY Study: TriVascular Evaluation of Females Who Are Underrepresented Candidates for Abdominal Aortic Aneurysm Repair
Brief Title: LUCY Study: TriVascular Evaluation of Females Who Are Underrepresented Candidates for Abdominal Aortic Aneurysm Repair
Acronym: LUCY
Status: Completed | Type: Observational
Sponsor: TriVascular, Inc. (Industry)
Responsible Party: Sponsor
Organization: Endologix (Industry)
Other Study IDs: 771-0016
Record Dates: First submitted 2015-06-18; First posted 2015-06-24 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal; Aortic; Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Female (Treatment Group): Device: Ovation Abdominal Stent Graft Platform
  Interventions: Device: Ovation Abdominal Stent Graft Platform
- Male (Control Group): Device: Ovation Abdominal Stent Graft Platform
  Interventions: Device: Ovation Abdominal Stent Graft Platform

INTERVENTIONS:
Device: Ovation Abdominal Stent Graft Platform

SUMMARY:
The LUCY Study is a prospective, consecutively enrolling, non-randomized multi center post-market registry to evaluate the low profile Ovation ® Abdominal Stent Graft Platform when used in the endovascular treatment of female patients.

DETAILED DESCRIPTION:
The LUCY Study is a prospective, consecutively enrolling, non-randomized multi center post-market registry to evaluate the Ovation Abdominal Stent Graft Platform when used in the endovascular treatment of female patients.

The primary endpoint is the Major Adverse Event (MAE) rate within 30 days of the initial procedure. MAEs will be adjudicated and reported based upon an independent Clinical Events Committee (CEC).

Secondary endpoints of the study will be achieved by demonstrating the benefits in female patients (Treatment Group) are comparable to male patients (Control Group) despite the fact that historically fewer female patients have been eligible for EVAR, and they have experienced a higher rate of access-related complications and higher mortality rates. Secondary endpoints will be evaluated through 1 year (365 ± 60 days) post-procedure.

A maximum of 45 sites across the United States are expected to enroll 225 subjects (75 females in the Treatment Group and 150 males in the Control Group).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > 18 years of age.
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study).
3. Patient has signed an Institutional Review Board (IRB) approved Informed Consent Form.
4. Patient is considered by the treating physician to be a candidate for elective open surgical repair of the AAA (i.e., category I, II, or III per American Society of Anesthesiology (ASA) classification; refer to Appendix II: ASA Classification System). ASA category IV patients may be enrolled provided their life expectancy is greater than 1 year.
5. Patient has an infrarenal abdominal aortic aneurysm that meets at least one of the following:

   1. Abdominal aortic aneurysm >5.0 cm in diameter;
   2. Aneurysm has increased in size by 0.5 cm in last 6 months; or
   3. Maximum diameter of aneurysm exceeds 1.5 times the transverse dimension of an adjacent non-aneurysmal aortic segment.
6. Patient has suitable anatomy that allows use of the TriVascular Ovation Abdominal Platform:

   1. Iliac or femoral arteries that allow endovascular access with the TriVascular Ovation Abdominal Platform.
   2. Proximal aortic neck landing zone with an inner wall diameter of no less than 16 mm and no greater than 30 mm at 13 mm below the inferior renal artery.
   3. Distal iliac artery landing zone length (seal zone) of ≥10 mm. The resultant repair should preserve patency in at least one hypogastric artery.
   4. Distal iliac artery landing zone an inner wall diameter of no less than 8 mm and no greater than 25 mm.
   5. Distance from the most distal renal artery to most superior internal iliac artery measurement is at least 130 mm.
   6. Aortic angle of ≤ 60 degrees if proximal neck length is ≥10 mm and ≤ 45 degrees if proximal neck length is <10 mm.
7. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria

1. Patient has a need for emergent surgery.
2. Patient has a dissecting aneurysm.
3. Patient has an acutely ruptured aneurysm.
4. Patient has an acute vascular injury.
5. Patient has had a previous repair of the abdominal aortic aneurysm or an iliac artery in intended treatment zone.
6. Patient has a known thoracic aortic aneurysm or dissection that will require treatment (surgery or endovascular intervention) within the study period.
7. Patient has a mycotic aneurysm or has an active systemic infection.
8. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina).
9. Patient has had a myocardial infarction (MI) and/or stroke (CVA) within the past 6 months.
10. Patient requires use of techniques (e.g. Chimney graft) that would cover the renal arteries.
11. Patient requires planned adjunctive devices (e.g. renal stents) to complete the procedure.
12. Patient has a major surgical or interventional procedure planned during or within ±30 days of the AAA repair.
13. Patient has history of connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndrome).
14. Patient has history of bleeding disorders or refuses blood transfusions.
15. Patient has dialysis dependent renal failure or baseline serum creatinine level >2.0 mg/dl
16. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
17. Patient has a known allergy or intolerance to polytetrafluoroethylene (PTFE), PEG-based polymers, fluorinated ethylene propylene (FEP) or nitinol.
18. Patient has a body habitus that would inhibit X-ray visualization of the aorta.
19. Patient has a limited life expectancy of less than 1 year.
20. Patient is currently participating in an investigational device or drug clinical trial.
21. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll male and female subjects 18 years of age and older that have an AAA and meet all other inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Major Adverse Event (MAE) | 1 month (30 ± 10 days)

SECONDARY OUTCOMES:
Serious and Non-Serious Adverse Events | 1 year (365 ± 60 days)
Access-related vascular complications | 1 year (365 ± 60 days)
Technical (deployment) success | 1 year (365 ± 60 days)
Freedom from Type I & III endoleaks | 1 year (365 ± 60 days)
Freedom from migration | 1 year (365 ± 60 days)
Freedom from aneurysm enlargement | 1 year (365 ± 60 days)
Freedom from AAA rupture | 1 year (365 ± 60 days)
Freedom from conversion to open repair | 1 year (365 ± 60 days)
Freedom from AAA related secondary interventions | 1 year (365 ± 60 days)
Freedom from mortality (all cause and AAA related) | 1 year (365 ± 60 days)
Clinical Utility, including: | 1 year (365 ± 60 days)
  Blood loss, including if transfusion required, Duration of procedure, Length of hospital and ICU (if required) stay, Anesthesia type

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ash, MD, Study Chair — Christie Clinic Vein & Vascular Center; Venita Chandra, MD, Study Chair — Stanford School of Medicine; Eva Rzucidlo, MD, Study Chair — Geisel School of Medicine, Dartmouth; Ageliki Vouyouka, MD, Study Chair — MOUNT SINAI HOSPITAL; Monica Hunter, MD, Study Chair — Ohio Heart and Vascular Center
Locations (1):
- Stanford University, Stanford, California, United States